CLINICAL TRIAL: NCT05077241
Title: Efficacy of Home Inspiratory Muscle Training in Post-covid-19 Patients: a Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Patri-cia Angelica de Miranda Silva Nogueira, Pesquisador principal, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1a2b3c4d5e6f
Record Dates: First submitted 2021-06-30; First posted 2021-10-14 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Covid19
Keywords: covid-19; respiratory muscle strength; spirometry
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group - inspiratory muscle training group with load (Experimental): Experimental group: Inspiratory muscle training with POWERbreathe® (POWERbreathe®, HaB Ltd, Southam, UK) with 30% of Pimax. with weekly load increment of 10% of the Pimax value. initial. The sessions will consist of 30 repetitions, twice a day, one in the morning and one in the afternoon, 7 consecutive days a week, for 6 weeks. Individuals will be instructed to perform a rapid contraction of the inspiratory muscles and sustain it for 2 seconds in each maneuver, and will have the possibility to rest every 3 repetitions of the TMI, for 30 seconds, to avoid muscle fatigue or any other complication.
  Interventions: Device: Inspiratory muscle training
- Control group - inspiratory muscle training group without load (Placebo Comparator): Subjects will use a IMT POWERbreathe® (POWERbreathe®, HaB Ltd, Southam, UK) device without any load and will receive the same guidelines as experimental group (The sessions will consist of 30 repetitions, twice a day, one in the morning and one in the afternoon, 7 consecutive days a week, for 6 weeks. Individuals will be instructed to perform a rapid contraction of the inspiratory muscles and sustain it for 2 seconds in each maneuver, and will have the possibility to rest every 3 repetitions of the TMI, for 30 seconds, to avoid muscle fatigue or any other complication). At the end of the research, the control group will have the right to experimental treatment with the IMT protocol, if this is effective.
  Interventions: Device: Inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — Individuals will be instructed to perform a rapid contraction of the inspiratory muscles against a load and sustain it for 2 seconds in each maneuver.

SUMMARY:
INTRODUCTION: Coronavirus 2019 disease (COVID-19), caused by the Severe Acute Respiratory Syndrome (SRAG) of coronavirus 2 (SARS-CoV-2) surpassed the global number of 119,603,761 cases, with more than 2,649,722 reported deaths . There is sufficient evidence for a possible post-covid-19 syndrome, designating sequelae with persistent symptoms. Respiratory muscle training improves respiratory muscle strength, exercise capacity, diaphragm muscle thickness, and dyspnea in various patient populations, especially in those with the greatest reduction in basal respiratory muscle strength. OBJECTIVE: To evaluate the effectiveness of a home inspiratory muscle training protocol in improving respiratory muscle strength, dyspnea and quality of life in post-Covid-19 patients. MATERIALS AND METHODS: This is a clinical, controlled, randomized and blind trial, which will be carried out at the Institute of Tropical Medicine of the Federal University of Rio Grande do Norte. The sample size will be performed using GPower software version 3.1.9.2 (Kiel, Germany) for Windows and will be established after conducting a pilot study with 5 participants in each group (total of 10 subjects) for a hypothetical two-way ANOVA test, using the main variable the Maximum Inspiratory Pressure (PImax.). The subjects included in the research will undergo three evaluation moments: Pre-training (Initial), Post-training (6 weeks) and Retention Test (24 weeks) for clinical evaluation form, anthropometric measures, respiratory muscle strength, volumes and capacities pulmonary symptoms, dyspnea, perceived exertion and fatigue, handgrip strength, six-minute walk test, anxiety and depression, post-covid functional status. After the initial assessment, all volunteers will receive a POWERbreathe® device (POWERbreathe®, HaB Ltd, Southam, UK) to carry out the training. EXPECTED RESULTS: provide a safe, effective and easy-to-perform treatment for post-covid-19 patients.

DETAILED DESCRIPTION:
The subjects included in the research will go through three evaluation moments: Pre-training (Initial), Post-training (3 and 6 weeks) and Retention Test (12 and 24 weeks).

After recruitment, participants will be invited to attend the Institute of Tropical Medicine to carry out an initial assessment by an evaluator previously trained and blinded to the intervention allocation group and will include anamnesis and physical examination, with measurement of vital signs, anthropometric measurements, assessment of lung volumes, respiratory muscle strength, peripheral muscle strength, quality of life, anxiety and depression, functional status and the 6-minute walk test.

After the initial evaluation, all volunteers will receive a POWERbreathe® device (POWERbreathe®, HaB Ltd, Southam, UK), to carry out the training, and will be individually instructed on how to use it and on the performance of the protocol. They will conduct an experimental session to familiarize themselves with the device that will not be considered for review. Every three days, volunteers will receive a phone call from researcher 2, who will not participate in the assessment, to confirm whether the exercise with the POWERbreathe® was being performed properly at the frequency and load set and if there were any doubts regarding the protocol. At the end of each week, participants will receive a video call from researcher 2 to adjust the device according to the weekly load progression of G1.

All evaluation moments (pre-training, post-training and retention test) will be performed by a single evaluator (Evaluator 1) - who will not know which group the subject will be allocated to - and recorded in the evaluation form developed for the project. A second researcher (Evaluator 2) will be responsible for applying the training protocols to the subjects.

ELIGIBILITY:
Inclusion Criteria:

* subjects of both sexes, sedentary, within two months of a diagnosis of COVID-19 confirmed by RT-PCR, aged over 18 years and without any underlying respiratory disease, with adequate cognitive status defined through the Mini Mental State Examination and reduced muscle strength respiratory, defined through the assessment of the maximum inspiratory pressure.

Exclusion Criteria:

* subjects who present any condition that makes it impossible to carry out the assessments and protocols, complications that justify the interruption of data collection, such as syncope, severe chest pain, coughing up blood, those who request withdrawal from the study and who present adverse effects such as hospitalization by exacerbation of the clinical picture.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | Change from baseline at 3 weeks, 6 weeks, 12 weeks and 24 weeks.
  The assessment of respiratory muscle strength will be performed by measuring the maximum respiratory pressures (Maximum Inspiratory Pressure: PImax and Maximum Expiratory Pressure: PEmax) through the use of an analog manometer (GERAR®, São Paulo, Brazil) with an operating range of ± 300 cmH2O and equipped with a mouthpiece adapter, containing an exhaust valve through an orifice of approximately 2mm in diameter to prevent the increase of intraoral pressure. For data analysis, at least three reproducible maneuvers will be used, with variability less than 20%, and the highest value will be recorded. The normality references for the calculation of maximal respiratory pressures as a function of age and gender will respect the description of the method used by Pessoa et al. (2014) for the Brazilian population.
Dyspnea - Medical Research Council | Change from baseline at 3 weeks, 6 weeks, 12 weeks and 24 weeks.
  Dyspnea will be assessed using the scale adapted to Portuguese by the Medical Research Council. The scale will allow the volunteer to indicate the extent to which their shortness of breath affected their mobility in daily activities. The scores range from 1 to 5, whose higher values refer to greater dyspnea, and the lower values reflect less dyspnea and will be chosen by the participant (BESTALL et al., 1999).
Quality of life (SF-36) | Change from baseline at 3 weeks, 6 weeks, 12 weeks and 24 weeks.
  The Medical Outcomes Study 36-Item Short Health Form Survey (SF-36) is a multidimensional questionnaire translated and validated for the Brazilian reality (CICONELLI et al., 1999; LAGUARDIA et al., 2011) that was developed to assess quality of life related to health. Scores range from 0 to 100 for each subscale, with higher scores being indicative of a better health-related quality of life (WARE; SHERBOURNE, 1992).

SECONDARY OUTCOMES:
Pulmonary function | Change from baseline at 3 weeks, 6 weeks, 12 weeks and 24 weeks.
  All participants will undergo an evaluation by a Koko Digidoser model spirometer (Spide, Longmont, USA) to verify lung volumes and capacities. At least three tests will be performed, with a variation of less than 5% and the highest value obtained in one of the tests will be compared with the predicted values of pulmonary function parameters for the Brazilian population. FEV1 and FVC will be assessed. The predicted values will be calculated using the reference values (PEREIRA et al., 2007).
Exercise tolerance | Change from baseline at 3 weeks, 6 weeks, 12 weeks and 24 weeks.
  The six-minute walk test assesses a submaximal level of functional capacity during exercise, measuring the distance a patient can walk on a flat surface of 30 meters for six minutes. At the end of the six minutes the number of laps will be registered and a marker placed on the floor beside the subject (ATS, 2002). The distance covered in the last lap will be measured by a tape measure and the total distance obtained by multiplying the number of laps by the measure of space and adding the distance covered in the last lap (ATS, 2002). The method to assess the predicted distance will follow the equations proposed in the literature, based on the gender, weight, age and height of the participants (ENRIGHT; SHERRILL, 1998).
Functional status | Change from baseline at 3 weeks, 6 weeks, 12 weeks and 24 weeks.
  The post-covid-19 functional status scale assesses relevant aspects of daily life during follow-up after infection. The scale contains six items ranging from zero to five and comprises the full range of functional outcomes with a focus on limitations of tasks and activities of daily living (home, work/study and lifestyle changes). The general classification corresponds to the worst functional status indicated by the patients' responses (the highest degree corresponding to the greatest limitations) (KLOK et al., 2020).
Anxiety and depression | Change from baseline at 3 weeks, 6 weeks, 12 weeks and 24 weeks.
  Depression Self-Rating Scales (SDS) and Anxiety Self-Rating Scale (SAS) will be explored to assess depression and anxiety in groups. Both the SDS and the SAS have 20 items, each of which will be scored on a scale of 1-4, and the higher the score, the more severe the degree of depression and anxiety (ZUNG, 1991).
Peripheral muscle strength | Change from baseline at 3 weeks, 6 weeks, 12 weeks and 24 weeks.
  The handgrip strength will be measured with the manual hydraulic dynamometer (Saehan®). It will be quantified by measuring the amount of maximum isometric force that the dominant hand can squeeze the dynamometer. The cut-off point will be <27kg for men and <16kg for women (CRUZ-JENTOFT et al., 2019).
Adverse effects and adherence | Change from baseline at 3 weeks, 6 weeks, 12 weeks and 24 weeks.
  For the assessment of adverse effects, a training diary will be provided to all study volunteers, in which all training days they must take will be provided and a blank space for positive and/or negative observations and to record any complications during and/or after training sessions. For analysis of adherence to training will be considered every time they mark the tables signaling the performance of the session. The sum of all sessions made will be carried out and these will be divided by the total number of sessions that the participants must do.
Physical activity level | Change from baseline at 3 weeks, 6 weeks, 12 weeks and 24 weeks.
  The level of physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ). The long version of the IPAQ (ANNEX 5), adapted (MAZO; BENEDETTI, 2001) and validated for the Brazilian population (BENEDETTI et al., 2008) comprises 5 domains and 15 questions. Participants will be classified as very active, active, irregularly active and sedentary (MATSUDO et al., 2002).
Cognition | baseline
  The Mini Mental State Examination (MMSE) will be used for cognitive screening in the elderly. It consists of two sections that assess cognitive functions. The final score is 30 points. Higher score values indicate greater cognitive performance (FOLSTEIN et al., 1975). The proposed cutoff scores will be used to minimize the influence of the level of education on the total scores (BERTOLUCCI et al., 1994).
Perception of effort and fatigue | Change from baseline at 3 weeks, 6 weeks, 12 weeks and 24 weeks.
  Individuals will be asked separately about their subjective perception of effort during breathing and fatigue in the lower limbs. To quantify it was the modified Borg RPE scale. The scale had numerical values from 0 to 10 and expressions that classify the degree of difficulty, whose higher values reflect a greater feeling of breathlessness (BORG, 2007).
Functional independence measure | Change from baseline at 3 weeks, 6 weeks, 12 weeks and 24 weeks.
  The FIM is a scale used to analyze the individual's performance to perform Basic Activities of Daily Living (ABVD) and Instrumental Activities of Daily Living (IADL) in a set of 18 tasks, related to the motor domains (self-care, sphincter control, transfers and locomotion). Thus, the total scale score ranges from eighteen points to one hundred and twenty-six points, with a classification of severe functional impairment (18-36 points), moderate (37-89 points), mild (90-126 points) (Riberto et al. 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia Angélica de Miranda Silva Nogueira., Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (2):
- Brazil (2):
  - Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte
  - Gabriely Azevêdo, Natal, Rio Grande do Norte

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goncalo Silva GA, Nogueira IDB, da Silva Chiappa GR, Nogueira PAMS. Efficacy of home-based inspiratory muscle training in patients post-covid-19: Protocol for a randomized clinical trial. PLoS One. 2023 May 4;18(5):e0279310. doi: 10.1371/journal.pone.0279310. eCollection 2023. PMID 37141260